CLINICAL TRIAL: NCT01507051
Title: Randomized, Placebo-controlled, Parallel-group Study in Healthy Male Subjects to Investigate the Pharmacodynamics During the Switching Procedure From Warfarin to Rivaroxaban
Brief Title: Switching Study From Warfarin to Rivaroxaban
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 10849; 2008-005540-16 (EudraCT Number)
Record Dates: First submitted 2011-12-05; First posted 2012-01-10 (Estimated); Results first posted 2012-04-26 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Venous Thrombosis
Keywords: Rivaroxaban; Xa-Factors; Warfarin; Thrombosis; Embolism
MeSH Terms: conditions — Venous Thrombosis; Thrombosis; Embolism | interventions — Warfarin; Rivaroxaban; Vitamin K; Vitamin K 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Warfarin followed by Rivaroxaban (Xarelto, BAY59-7939) (Experimental): Days -6 and -5: 10 mg warfarin once daily or lower depending on international normalized ratio (INR); Days -4 to -1 (could be prolonged by two days): 2.5, 5, 10, 12.5 or 15 mg warfarin once daily depending on INR; Days 0 to 3: 20 mg rivaroxaban once daily; Day 5: 10 mg vitamin K once daily
  Interventions: Drug: Warfarin (Coumadin); Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Vitamin K (Konakion)
- Warfarin followed by Placebo (Placebo Comparator): Days -6 and -5: 10 mg warfarin once daily or lower depending on INR; Days -4 to -1 (could be prolonged by two days): 2.5, 5, 10, 12.5 or 15 mg warfarin once daily depending on INR; Days 0 to 3: 1 tablet matching placebo once daily; Day 5: 10 mg vitamin K once daily
  Interventions: Drug: Warfarin (Coumadin); Drug: Placebo; Drug: Vitamin K (Konakion)
- Rivaroxaban (Xarelto, BAY59-7939) (Active Comparator): Days 0 to 3: 20 mg rivaroxaban once daily
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Warfarin (Coumadin) — Days -6 and -5: 10 mg warfarin (Coumadin) once daily, dosage lower if the INR is already high on day -5; Days -4 to -1 (could be prolonged by two days): 2.5, 5, 10, 12.5 or 15 mg warfarin (Coumadin) once daily, dosage depending on INR
  Arms: Warfarin followed by Placebo; Warfarin followed by Rivaroxaban (Xarelto, BAY59-7939)
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Days 0 to 3: 20 mg rivaroxaban once daily
  Arms: Rivaroxaban (Xarelto, BAY59-7939); Warfarin followed by Rivaroxaban (Xarelto, BAY59-7939)
Drug: Placebo — Days 0 to 3: 1 tablet placebo, identical to active tablet
  Arms: Warfarin followed by Placebo
Drug: Vitamin K (Konakion) — Day 5: 10 mg vitamin K (Konakion) once daily
  Arms: Warfarin followed by Placebo; Warfarin followed by Rivaroxaban (Xarelto, BAY59-7939)

SUMMARY:
The study objective is to investigate the pharmacodynamics (effects of a drug product) when switching the treatment from warfarin to rivaroxaban.

84 young, healthy subjects will participate; they will be treated following a randomized, parallel-group (Treatments A, B, and C), placebo-controlled (Treatment B), and single-blind (Treatments A and B) design.

The first two groups (A, B) will receive warfarin for approximately one week to adjust their blood coagulation values to a specific level, i.e. to maintain an INR (international normalized ratio) of 2.0 - 3.0. This range is commonly used for long-term anticoagulant treatment.

The first group (A) will receive rivaroxaban for four days, the second group (B) will take placebo. On the last day, all subjects in groups A and B will receive vitamin K to neutralize the effects of warfarin. The third group (C) will not undergo prior treatment with warfarin but will receive rivaroxaban for four days.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years of age;
* Normal body weight: BMI (body mass index) between 18 and 29 kg/m2;
* Pharmacogenetics: subjects who are homozygous for the wildtype allele 2C9*1 and who are carriers of the C-allele at positions 6484 and 7566 of the VKORC1 (vitamin K epoxide reductase) gene, respectively

Exclusion Criteria:

* Relevant deviation from the normal range in the clinical examination;
* Relevant deviation from the normal range in clinical chemistry, hematology or urinalysis;
* Resting heart rate in the awake subject below 45 BPM (beats per minute) or above 90 BPM;
* Systolic blood pressure below 100 mmHg or above 140 mmHg; and Diastolic blood pressure above 85 mmHg;
* Relevant pathological changes in the ECG (electrocardiogram) such as a second or third-degree AV block, prolongation of the QRS (QRS complex in ECG) complex over 120 msec or of the QT / QTc-interval over 450 msec (QT interval in ECG, QTc interval corrected for heart rate);
* Subject is tested to be HIV-1/2Ab, p24Ag, HbsAg or HCV-Ab positive;
* Known coagulation disorders (e.g. von Willebrand's disease, haemophiliac);
* Known disorders with increased bleeding risks (e.g. periodontosis, hemorrhoids, acute gastritis, peptic ulcer);
* Known sensitivity to common causes of bleeding (e.g. nasal);
* Recent or planned surgical or diagnostic procedures at the central nervous system (CNS) or eye;
* Subjects with hyperlipidemia (Coumadin / warfarin warning)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - Cologne, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia

REFERENCES:
- [Result] Kubitza D, Becka M, Muck W, Kratzschmar J. Pharmacodynamics and pharmacokinetics during the transition from warfarin to rivaroxaban: a randomized study in healthy subjects. Br J Clin Pharmacol. 2014 Aug;78(2):353-63. doi: 10.1111/bcp.12349. PMID 24528331
- See also: Click here and search for results posted for EMA — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by 2 centers in Germany: ClinPharmCologne - MEDA Manufacturing GmbH, Neurather Ring 1, 51063 Koeln, and CRS Clinical-Research-Services Moenchengladbach GmbH, Hindenburgstrasse 304-306, 41061 Moenchengladbach. 84 participants were planned to participate (n=28 per group; minimum completion target n=75, n=25 per group).
Pre-assignment Details: 488 participants were screened, 392 were dropped. 96 participants were included in the study, 55 by Trial Unit 1 ClinPharmCologne, and 41 by Trial Unit 2 CRS Moenchengladbach. 91 participants were included in the safety set, 84 participants were valid for the assessment of pharmacokinetics and pharmacodynamics (PK/PD set).
Groups:
- Group A: Warfarin Followed by Rivaroxaban: Days -6 and -5: 10 mg warfarin once daily or lower depending on INR; Days -4 to -1 (could be prolonged by two days): 2.5, 5, 10, 12.5 or 15 mg warfarin once daily depending on INR; Days 0 to 3: 20 mg rivaroxaban once daily; Day 5: 10 mg vitamin K once daily
- Group B: Warfarin Followed by Placebo: Days -6 and -5: 10 mg warfarin once daily or lower depending on INR; Days -4 to -1 (could be prolonged by two days): 2.5, 5, 10, 12.5 or 15 mg warfarin once daily depending on INR; Days 0 to 3: 1 tablet matching placebo once daily; Day 5: 10 mg vitamin K once daily
- Group C: Rivaroxaban Without Any Pre-treatment With Warfarin: Days 0 to 3: 20 mg rivaroxaban once daily
- Group D: Warfarin Alone: Days -6 to -1 (could be prolonged by 2 days): dose 15 mg to 2.5 mg, dosing depending on INR
Period: Overall Study
Arm/Group | Group A: Warfarin Followed by Rivaroxaban | Group B: Warfarin Followed by Placebo | Group C: Rivaroxaban Without Any Pre-treatment With Warfarin | Group D: Warfarin Alone
Started | 29 | 31 | 29 | 7
Warfarin run-in Phase | 28 | 28 | 0 | 7 (Safety Population: in RG4)
Received Placebo or Rivaroxaban | 28 (Safety Population: in RG1 and in RG4 (RG = Reporting Group for Safety Data)) | 28 (Safety Population: in RG2 and in RG4) | 28 (Safety Population: in RG3) | 0
Completed | 27 | 28 | 28 | 0
Not Completed | 2 | 3 | 1 | 7
Not completed — Withdrawal by Subject | 1 | 3 | 1 | 6
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939): Days -6 and -5: 10 mg warfarin once daily or lower depending on INR; Days -4 to -1 (could be prolonged by two days): 2.5, 5, 10, 12.5 or 15 mg warfarin once daily depending on INR; Days 0 to 3: 20 mg rivaroxaban once daily; Day 5: 10 mg vitamin K once daily
- Warfarin Alone: Days -6 to -1 (could be prolonged by 2 days): dose 15 mg to 2.5 mg, dosing depending on INR
- Total: Total of all reporting groups
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Alone | Total
Number analyzed (Participants) | 28 | 28 | 28 | 7 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (7.2) | 30.7 (7.5) | 34.8 (8.0) | 34.6 (6.9) | 32.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 28 | 28 | 28 | 7 | 91

OUTCOME MEASURES:

1. Primary Outcome: Emax (Maximum Effect) on Prothrombin Time (PT) (Coagulation Test)
Description: Prothrombin time (PT) is a global clotting test assessing the extrinsic pathway of the blood coagulation cascade. The test is sensitive for deficiencies of Factors II, V, VII, and X, with sensitivity being best for Factors V, VII, and X and less pronounced for Factor II. The initial read-out is in seconds. Higher values than the baseline indicate anticoagulant effects. Emax on PT was measured as the ratio of maximum PT (measured in seconds) divided by PT (measured in seconds) at baseline.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio | 4.393 (18.03) | 1.884 (10.35) | 1.573 (9.98)
Statistical Analysis 1: Comparison: Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) vs Rivaroxaban (Xarelto, BAY59-7939); Test type: Superiority or Other; p < 0.0001, ANOVA; Geometric LS-Mean Ratio = 2.793, 90% CI [2.633 to 2.962]

2. Primary Outcome: Emax,BA (Baseline Adjusted Maximum Effect) on Prothrombin Time (Coagulation Test)
Description: Prothrombin time (PT) is a global clotting test assessing the extrinsic pathway of the blood coagulation cascade. The test is sensitive for deficiencies of Factors II, V, VII, and X, with sensitivity being best for Factors V, VII, and X and less pronounced for Factor II. The initial read-out is in seconds. Higher values than the baseline indicate anticoagulant effects. Emax,BA on PT was measured as maximum PT (measured in seconds) minus PT (measured in seconds) at baseline.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: seconds
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
seconds | 44.98 (20.84) | 11.59 (19.52) | 7.31 (23.72)
Statistical Analysis 1: Comparison: Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) vs Rivaroxaban (Xarelto, BAY59-7939); Test type: Superiority or Other; p < 0.0001, ANOVA; Geometric LS-Mean Ratio = 6.151, 90% CI [5.598 to 6.759]

3. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of Prothrombin Time (Coagulation Test)
Description: Prothrombin time (PT) is a global clotting test assessing the extrinsic pathway of the blood coagulation cascade. The test is sensitive for deficiencies of Factors II, V, VII, and X, with sensitivity being best for Factors V, VII, and X and less pronounced for Factor II. The initial read-out is in seconds. Higher values than the baseline indicate anticoagulant effects. AUC(0-tn) of PT was the area under the measurement (PT [measured in seconds] at different time-points divided by PT [measured in seconds] at baseline) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio*h | 55.36 (13.36) | 37.89 (9.92) | 20.41 (33.52)

4. Secondary Outcome: AUCBA(0-tn) (Baseline Adjusted Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of Prothrombin Time (Coagulation Test)
Description: Prothrombin time (PT) is a global clotting test assessing the extrinsic pathway of the blood coagulation cascade. The test is sensitive for deficiencies of Factors II, V, VII, and X, with sensitivity being best for Factors V, VII, and X and less pronounced for Factor II. The initial read-out is in seconds. Higher values than the baseline indicate anticoagulant effects. AUCBA(0-tn) of PT was the area under the measurement (PT [measured in seconds] at different time-points minus PT [measured in seconds] at baseline) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: s*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
s*h | 413.4 (19.87) | 179.9 (26.58) | 33.06 (55.70)

5. Secondary Outcome: Emax on PT (Measured as INR=International Normalized Ratio)
Description: Prothrombin time - INR measured in seconds that is calculated as INR which is a correction for PT assay differences and an optimization to measure vitamin K antagonists. Higher values than the baseline indicate anticoagulant effects. Emax on PT (INR) was measured as the ratio of maximum INR divided by baseline INR.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio | 6.655 (23.39) | 2.250 (13.19) | 1.793 (12.87)

6. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) for PT (Measured as INR=International Normalized Ratio)
Description: Prothrombin time - INR measured in seconds that is calculated as INR which is a correction for PT assay differences and an optimization to measure vitamin K antagonists. Higher values than the baseline indicate anticoagulant effects. AUC(0-tn) of PT (INR) was the area under the measurement (PT measured as INR at different time-points divided by PT measured as INR at baseline) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio*h | 72.30 (17.35) | 43.60 (12.81) | 23.21 (30.63)

7. Secondary Outcome: Emax on Factor Xa Activity
Description: Test to measure the activity of endogenous Factor Xa. Emax on Factor Xa activity was calculated as 100*(Factor Xa activity at baseline [measured as activity per mL] - minimum of Factor Xa activity [measured as activity per mL]) / Factor Xa activity at baseline [measured as activity per mL].
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of inhibition
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
Percentage of inhibition | 75.95 (6.56) | 43.41 (12.67) | 49.73 (13.86)

8. Secondary Outcome: AUC(0-tn) (Area Under the Inverse Measurement Versus Time Curve From Time 0 to the Last Data Point) of Factor Xa Activity
Description: Test to measure the activity of endogenous Factor Xa. AUC(0-tn) of Factor Xa activity was the area under the inverse measurement [100*(Factor Xa activity at baseline (measured as activity per mL) - Factor Xa activity (measured as activity per mL) at different time-points) / Factor Xa activity at baseline (measured as activity per mL)] versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of inhibition*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
Percentage of inhibition*h | 1238 (12.28) | 834.8 (19.44) | 514.1 (27.90)

9. Secondary Outcome: Emax (Maximum Effect) on Anti-Factor Xa Activity
Description: This is a method for measuring the inhibition of Factor Xa activity determined by an ex vivo using a photometric method. Higher Values than the baseline indicate a more pronounced inhibition. Emax on anti-Factor Xa activity was measured as the ratio of maximum anti-Factor Xa activity (measured in U/L) divided by anti-Factor Xa activity (measured in U/L) at baseline.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set; derived parameter could not be evaluated for all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 12 | 27
ratio | 15.83 (56.06) | 2.281 (112.7) | 18.57 (42.99)

10. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of Anti-Factor Xa Activity
Description: This is a method for measuring the inhibition of Factor Xa activity determined by an ex vivo using a photometric method. Higher Values than the baseline indicate a more pronounced inhibition. AUC(0-tn) of anti-Factor Xa activity was the area under the measurement (anti-Factor Xa activity [measured in U/L] at different time-points divided by anti-Factor Xa activity [measured in U/L] at baseline) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set; derived parameter could not be evaluated for all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 12 | 27
ratio*h | 124.9 (68.84) | 19.63 (202.0) | 151.6 (38.88)

11. Secondary Outcome: Emax (Maximum Effect) on aPTT (Activated Partial Thromboplastin Time)
Description: The aPTT is a screening test for the intrinsic pathway and is sensitive for deficiencies of Factors I, II, V, VIII, IX, X, XI and XII. Higher values than the baseline indicate anticoagulant effects. Emax on aPTT was measured as the ratio of maximum aPTT (measured in seconds) divided by aPTT (measured in seconds) at baseline.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio | 1.843 (10.55) | 1.304 (15.07) | 1.409 (6.19)

12. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of aPTT (Activated Partial Thromboplastin Time)
Description: The aPTT is a screening test for the intrinsic pathway and is sensitive for deficiencies of Factors I, II, V, VIII, IX, X, XI and XII. Higher values than the baseline indicate anticoagulant effects. AUC(0-tn) of aPTT was the area under the measurement (aPTT [measured in seconds] at different time-points divided by aPTT [measured in seconds] at baseline) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio*h | 32.48 (9.41) | 22.55 (56.41) | 21.82 (42.67)

13. Secondary Outcome: Emax (Maximum Effect) on HepTest (Coagulation Test)
Description: This coagulation test was developed to monitor heparin and especially low-molecular weight heparins (LMWH). It is sensitive to measure Factor X. Higher values than the baseline indicate anticoagulant effects. Emax on HepTest was measured as the ratio of maximum HepTest (measured in seconds) divided by HepTest (measured in seconds) at baseline.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set; derived parameter could not be evaluated for all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 23 | 28
ratio | 2.148 (14.20) | 1.163 (19.78) | 2.009 (12.13)

14. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of HepTest (Coagulation Test)
Description: This coagulation test was developed to monitor heparin and especially low-molecular weight heparins (LMWH). It is sensitive to measure Factor X. Higher values than the baseline indicate anticoagulant effects. AUC(0-tn) of HepTest was the area under the measurement (HepTest [measured in seconds] at different time-points divided by HepTest [measured in seconds] at baseline) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set; derived parameter could not be evaluated for all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 20 | 28
ratio*h | 27.37 (32.90) | 15.08 (125.9) | 28.25 (29.31)

15. Secondary Outcome: Emax (Maximum Effect) on PiCT (Prothrombinase-induced Clotting Time)
Description: This coagulation test can be adapted to measure different anticoagulants, including inhibitors of Factor X. Higher values than the baseline indicate anticoagulant effects. Emax on PiCT was measured as the ratio of maximum PiCT (measured in seconds) divided by PiCT (measured in seconds) at baseline.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set; derived parameter could not be evaluated for all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 18 | 27
ratio | 3.158 (27.20) | 1.139 (21.36) | 2.723 (20.69)

16. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of PiCT (Prothrombinase-induced Clotting Time)
Description: This coagulation test can be adapted to measure different anticoagulants, including inhibitors of Factor X. Higher values than the baseline indicate anticoagulant effects. AUC(0-tn) of PiCT was the area under the measurement (PiCT [measured in seconds] at different time-points divided by PiCT [measured in seconds] at baseline) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set; derived parameter could not be evaluated for all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 12 | 26
ratio*h | 37.36 (38.40) | 4.221 (429.5) | 39.20 (8.91)

17. Secondary Outcome: Emax (Maximum Effect) on ETP (Endogenous Thrombin Potential) AUC
Description: ETP AUC assesses the overall function of the clotting cascade. The AUC assesses the overall ability to generate thrombin. Decreasing values compared to baseline indicate an anticoagulant effect. Emax on ETP AUC was measured as the ratio of ETP AUC (measured in nm*min as integral of fluorescence measurements) at baseline divided by minimum ETP AUC (measured in nm*min as integral of fluorescence measurements).
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio | 4.257 (24.41) | 2.610 (22.05) | 1.813 (25.45)

18. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of ETP (Endogenous Thrombin Potential) AUC
Description: ETP AUC assesses the overall function of the clotting cascade. The AUC assesses the overall ability to generate thrombin. Decreasing values compared to baseline indicate an anticoagulant effect. AUC(0-tn) of ETP AUC was the area under the measurement (ETP AUC [measured in nm*min as integral of fluorescence measurements] at baseline divided by ETP AUC [measured in nm*min as integral of fluorescence measurements] at different time-points) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio*h | 69.69 (25.83) | 51.28 (17.90) | 18.06 (78.12)

19. Secondary Outcome: Emax (Maximum Effect) on ETP (Endogenous Thrombin Potential) Lag Time
Description: ETP lag time assesses the overall function of the clotting cascade. The lag time assesses the time required until thrombin is generated. Increasing values compared to baseline indicate an anticoagulant effect. Emax on ETP lag time was measured as the ratio of maximum ETP lag time (in minutes as measure for the start of coagulation) divided by ETP lag time (in minutes as measure for the start of coagulation) at baseline.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio | 3.954 (19.02) | 1.748 (18.49) | 2.569 (9.83)

20. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of ETP (Endogenous Thrombin Potential) Lag Time
Description: ETP lag time assesses the overall function of the clotting cascade. The lag time assesses the time required until thrombin is generated. Increasing values compared to baseline indicate an anticoagulant effect. AUC(0-tn) of ETP lag time was the area under the measurement (ETP lag time [in minutes as measure for the start of coagulation] at different time-points divided by ETP lag time [in minutes as measure for the start of coagulation] at baseline) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio*h | 63.75 (17.88) | 34.93 (20.83) | 42.79 (9.54)

21. Secondary Outcome: Emax (Maximum Effect) on ETP (Endogenous Thrombin Potential) Peak
Description: ETP peak assesses the overall function of the clotting cascade. The peak assesses the overall maximal ability to generate thrombin. Decreasing values compared to baseline indicate an anticoagulant effect. Emax on ETP peak was measured as the ratio of ETP peak (measured in nm as maximum coagulation activity) at baseline divided by minimum ETP peak (measured in nm as maximum coagulation activity).
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio | 18.73 (44.08) | 2.523 (44.17) | 6.758 (33.31)

22. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of ETP (Endogenous Thrombin Potential) Peak
Description: ETP peak assesses the overall function of the clotting cascade. The peak assesses the overall maximal ability to generate thrombin. Decreasing values compared to baseline indicate an anticoagulant effect. AUC(0-tn) of ETP peak was the area under the measurement (ETP peak [measured in nm as maximum coagulation activity] at baseline divided by ETP peak measured [in nm as maximum coagulation activity] at different time-points) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio*h | 166.8 (45.97) | 46.75 (19.22) | 74.67 (27.40)

23. Secondary Outcome: Emax (Maximum Effect) on ETP (Endogenous Thrombin Potential) Peak Time
Description: ETP peak time assesses the overall function of the clotting cascade. The peak time assesses the time required to reach the maximal thrombin generation. Increasing values compared to baseline indicate an anticoagulant effect. Emax on ETP peak time was measured as the ratio of maximum ETP peak time (measured in minutes as time to reach the maximum coagulation activity) divided by ETP peak time (measured in minutes as time to reach the maximum coagulation activity) at baseline.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio | 4.164 (33.95) | 1.375 (20.87) | 3.790 (15.75)

24. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of ETP (Endogenous Thrombin Potential) Peak Time
Description: ETP peak time assesses the overall function of the clotting cascade. The peak time assesses the time required to reach the maximal thrombin generation. Increasing values compared to baseline indicate an anticoagulant effect. AUC(0-tn) of ETP peak time was the area under the measurement (ETP peak time [measured in minutes as time to reach the maximum coagulation activity] at different time-points divided by ETP peak time [measured in minutes as time to reach the maximum coagulation activity] at baseline) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio*h | 49.14 (28.10) | 19.83 (143.9) | 55.58 (12.47)

25. Secondary Outcome: Emax (Maximum Effect) on Factor VIIa Activity
Description: Factor VII is a coagulation factor that is required for the coagulation process. Emax on Factor VIIa activity was measured as the ratio of Factor VIIa activity (measured as percent of actual Factor VIIa activity compared to Factor VIIa activity in reference plasma) at baseline divided by minimum Factor VIIa activity (measured as percent of actual Factor VIIa activity compared to Factor VIIa activity in reference plasma).
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio | 12.80 (47.88) | 6.769 (53.51) | 1.346 (7.51)

26. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of Factor VIIa Activity
Description: Factor VII is a coagulation factor that is required for the coagulation process. AUC(0-tn) of Factor VIIa activity was the area under the measurement (Factor VIIa activity [measured as percent of actual Factor VIIa activity compared to Factor VIIa activity in reference plasma] at baseline divided by Factor VIIa activity [measured as percent of actual Factor VIIa activity compared to Factor VIIa activity in reference plasma] at different time-points) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio*h | 134.2 (44.70) | 94.83 (41.07) | 9.283 (70.62)

27. Secondary Outcome: Emax (Maximum Effect) on Factor IIa Activity
Description: Factor II (Thrombin) is a coagulation factor that is required for the coagulation process. Emax on Factor IIa activity was measured as the ratio of Factor IIa activity (measured as percent of actual Factor IIa activity compared to Factor IIa activity in reference plasma) at baseline divided by minimum Factor IIa activity (measured as percent of actual Factor IIa activity compared to Factor IIa activity in reference plasma).
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 28
ratio | 3.166 (16.09) | 2.958 (12.31) | 1.126 (5.08)

28. Secondary Outcome: AUC(0-tn) (Area Under the Measurement Versus Time Curve From Time 0 to the Last Data Point) of Factor IIa Activity
Description: Factor II (Thrombin) is a coagulation factor that is required for the coagulation process. AUC(0-tn) of Factor IIa activity was the area under the measurement (Factor IIa activity [measured as percent of actual Factor IIa activity compared to Factor IIa activity in reference plasma] at baseline divided by Factor IIa activity [measured as percent of actual Factor IIa activity compared to Factor IIa activity in reference plasma] at different time-points) versus time curve from time 0 to the last data point.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban or placebo
Population: PK/PD set; derived parameter could not be evaluated for all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio*h
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28 | 26
ratio*h | 62.26 (18.20) | 58.60 (15.18) | 3.908 (117.7)

29. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hours [AUC(0-24)] of Rivaroxaban After First Dose
Description: The AUC is a measure of systemic drug exposure which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample ([AUC(0-24)] is defined as area under the concentration vs. time curve from zero to 24 hours after first (single) dose).
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microg*h/L
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28
microg*h/L | 1639 (29.46) | 1722 (26.19)
Statistical Analysis 1: Comparison: Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) vs Rivaroxaban (Xarelto, BAY59-7939); Test type: Superiority or Other; p = 0.5008, ANOVA; Geometric LS-Mean Ratio (%) = 95.17, 95% CI [82.20 to 110.2]

30. Secondary Outcome: Maximum Drug Concentration in Plasma (Cmax) of Rivaroxaban After First Dose
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microg/L
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28
microg/L | 219.8 (30.94) | 221.0 (26.65)
Statistical Analysis 1: Comparison: Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) vs Rivaroxaban (Xarelto, BAY59-7939); Test type: Superiority or Other; p = 0.9429, ANOVA; Geometric LS-Mean Ratio (%) = 99.46, 95% CI [85.47 to 115.7]

31. Secondary Outcome: Half Life Associated With Terminal Slope (t1/2) of R-warfarin After the Last Dose of Warfarin
Description: Half-life refers to the elimination of the drug, i.e. the time it takes for the blood plasma concentration to reach half the concentration in the terminal phase of elimination.
Time Frame: Blood samples taken at 24, 30, 48, 54, 72, 96, and 120 h after the last administration of warfarin
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo
Number analyzed (Participants) | 28 | 28
hours | 40.08 (19.63) | 40.24 (29.43)
Statistical Analysis 1: Comparison: Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin Followed by Placebo; Test type: Superiority or Other; p = 0.9525, ANOVA; Geometric LS-Mean Ratio (%) = 100.4, 95% CI [88.00 to 114.5]

32. Secondary Outcome: Half Life Associated With Terminal Slope (t1/2) of S-warfarin After the Last Dose of Warfarin
Description: as for outcome 31
Time Frame: Blood samples taken at 24, 30, 48, 54, 72, 96, and 120 h after the last administration of warfarin
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo
Number analyzed (Participants) | 28 | 28
hours | 28.24 (17.95) | 27.08 (22.79)
Statistical Analysis 1: Comparison: Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) vs Warfarin Followed by Placebo; Test type: Superiority or Other; p = 0.4397, ANOVA; Geometric LS-Mean Ratio (%) = 95.87, 95% CI [85.99 to 106.9]

33. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hours Divided by Dose Per kg Body Weight [AUC(0-24)Norm] of Rivaroxaban After First Dose
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample; [AUC(0-24)norm] is defined as AUC divided by dose per kg body weight from zero to 24 hours after first (single) dose.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Kg*h/L
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28
Kg*h/L | 6.569 (27.55) | 6.901 (31.63)

34. Secondary Outcome: Maximum Drug Concentration in Plasma Divided by Dose Per kg Body Weight (Cmax,Norm) of Rivaroxaban After First Dose
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample; Cmax,norm is defined as Cmax divided by dose (mg) per kg body weight.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Kg/L
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28
Kg/L | 0.8812 (27.83) | 0.8857 (31.79)

35. Secondary Outcome: Time to Reach Maximum Drug Concentration in Plasma (Tmax) of Rivaroxaban After First Dose
Description: Tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban
Population: PK/PD set
Measure: Median (Full Range); unit: hours
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28
hours | 3.008 [1.000 to 4.000] | 3.000 [1.000 to 4.067]

36. Secondary Outcome: Drug Concentration in Plasma at Expected Time of Maximum (Peak) Concentration (Cpeak) of Rivaroxaban After Second to Fourth Dose
Description: Cpeak refers to the time after dosing when the drug concentration is expected to reach its maximum (peak) concentration.
Time Frame: Always 3 h after second, third, and fourth dose
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microg/L
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28
Microg/L
  second dose | 211.2 (28.72) | 206.7 (35.62)
  third dose | 206.1 (30.66) | 201.0 (30.65)
  fourth dose | 201.4 (77.43) | 214.5 (27.35)

37. Secondary Outcome: Drug Concentration in Plasma at Expected Time of Minimum (Trough) Concentration (Ctrough) of Rivaroxaban After Second to Fourth Dose
Description: Ctrough refers to the time after dosing when the drug concentration is expected to reach its minimum (trough) concentration.
Time Frame: Always 24 h after the second, third, and fourth dose
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microg/L
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 28 | 28
Microg/L
  second dose | 13.06 (50.64) | 17.07 (45.32)
  third dose | 14.34 (54.05) | 15.85 (47.92)
  fourth dose | 12.43 (85.96) | 15.61 (51.52)

38. Secondary Outcome: Half Life Associated With Terminal Slope (t1/2) of Rivaroxaban After Last Dose
Description: as for outcome 31
Time Frame: 3, 24, 48, and 72 h after the last administration of rivaroxaban
Population: PK/PD set; derived parameter could not be evaluated for all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 27 | 28
hours | 6.885 (42.48) | 6.931 (36.70)

39. Secondary Outcome: Drug Concentration in Plasma at Steady State at Expected Time of Minimum (Trough) Concentration (Ctrough,ss) of R-warfarin After the Last Dose of Warfarin
Description: Ctrough,ss refers to the drug concentration at steady state at the time when it is expected to reach its minimum (trough) concentration.
Time Frame: 0 h (predose) and 24 h after the last administration of warfarin
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microg/L
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo
Number analyzed (Participants) | 28 | 28
Microg/L
  before last administration | 754.4 (32.70) | 721.8 (25.56)
  after last administration | 740.2 (25.88) | 702.8 (28.39)

40. Secondary Outcome: Drug Concentration in Plasma at Steady State at Expected Time of Minimum (Trough) Concentration, Normalized by Dose (Ctrough,ss/D) of R-warfarin After the Last Dose of Warfarin
Description: Ctrough,ss/D refers to the drug concentration at steady state at the time when it is expected to reach its minimum (trough) concentration, normalized by dose.
Time Frame: 0 h (predose) and 24 h after the last administration of warfarin
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/Liter
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo
Number analyzed (Participants) | 28 | 28
1/Liter
  before last administration | 0.07154 (40.86) | 0.07843 (48.55)
  after last administration | 0.08633 (44.10) | 0.07915 (46.50)

41. Secondary Outcome: Drug Concentration in Plasma at Steady State at Expected Time of Minimum (Trough) Concentration (Ctrough,ss) of S-warfarin After the Last Dose of Warfarin
Description: as for outcome 39
Time Frame: 0 h (predose) and 24 h after the last administration of warfarin
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microg/L
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo
Number analyzed (Participants) | 28 | 28
Microg/L
  before last administration | 498.2 (38.93) | 429.9 (31.14)
  after last administration | 478.4 (26.17) | 424.9 (29.78)

42. Secondary Outcome: Drug Concentration in Plasma at Steady State at Expected Time of Minimum (Trough) Concentration, Normalized by Dose (Ctrough,ss/D) of S-warfarin After the Last Dose of Warfarin
Description: as for outcome 40
Time Frame: 0 h (predose) and 24 h after the last administration of warfarin
Population: PK/PD set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/Liter
Arm/Group | Warfarin Followed by Rivaroxaban (Xarelto, BAY59-7939) | Warfarin Followed by Placebo
Number analyzed (Participants) | 28 | 28
1/Liter
  before last administration | 0.04724 (43.96) | 0.04671 (53.03)
  after last administration | 0.05580 (43.11) | 0.04786 (38.96)

ADVERSE EVENTS:
Groups:
- RG1: Warfarin Followed by Rivaroxaban: All participants received warfarin and later rivaroxaban. Days -6 and -5: 10 mg warfarin once daily or lower depending on INR; Days -4 to -1 (could be prolonged by two days): 2.5, 5, 10, 12.5 or 15 mg warfarin once daily depending on INR; Days 0 to 3: 20 mg rivaroxaban once daily; Day 5: 10 mg vitamin K once daily. Note: Safety Data presented here include participants listed in Group A of the Participant Flow section.
- RG2: Warfarin Followed by Placebo: All participants received warfarin and later placebo. Days -6 and -5: 10 mg warfarin once daily or lower depending on INR; Days -4 to -1 (could be prolonged by two days): 2.5, 5, 10, 12.5 or 15 mg warfarin once daily depending on INR; Days 0 to 3: 1 tablet matching placebo once daily; Day 5: 10 mg vitamin K once daily. Note: Safety Data presented here include participants listed in Group B of the Participant Flow section.
- RG3: Rivaroxaban: All participants received rivaroxaban. Days 0 to 3: 20 mg rivaroxaban once daily. Note: Safety Data presented here include participants listed in Group C of the Participant Flow section.
- RG4: Warfarin Alone: All participants received warfarin in the Run-In Phase, who either received rivaroxaban or placebo afterwards, or discontinued the study. Days -6 to -1(could be prolonged by 2 days): dose 15 mg to 2.5 mg, dosing depending on INR. Note: Safety Data presented here include participants listed in Groups A, B (warfarin run-in only) and D of the Participant Flow section.
Arm/Group | RG1: Warfarin Followed by Rivaroxaban | RG2: Warfarin Followed by Placebo | RG3: Rivaroxaban | RG4: Warfarin Alone
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/63
Other Adverse Events (participants affected / at risk) | 14/28 | 12/28 | 10/28 | 21/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RG1: Warfarin Followed by Rivaroxaban (N=28) | RG2: Warfarin Followed by Placebo (N=28) | RG3: Rivaroxaban (N=28) | RG4: Warfarin Alone (N=63)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Urine output increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spontaneous penile erection (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any disclosure of study results by the Principal Investigator or investigators has to be in agreement with the sponsor.